CLINICAL TRIAL: NCT06243289
Title: Improving KIdney ¬Transplantation with Cellular Therapy Study
Brief Title: Improving KIdney Transplantation with Cellular Therapy Study
Acronym: i-KITCaT
Status: Terminated | Type: Observational
Why Stopped: Low recruitment
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Jennifer Li, CPI, Nephrologist and Transplant Physician, Western Sydney Local Health District
Other Study IDs: ikitcat
Record Dates: First submitted 2024-01-28; First posted 2024-02-06 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-02

CONDITIONS: Immune Tolerance; Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood collected for PBMC and DNA. DNA will be bio-banked for future renal related research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy participants: Volunteers with no kidney disease, autoimmune disease or major cardiovascular comorbidities
  Interventions: Other: Tolerance induction
- Participants with kidney disease: Includes patient with chronic kidney disease, dialysis or functioning transplant
  Interventions: Other: Tolerance induction

INTERVENTIONS:
Other: Tolerance induction — Exposure of peripheral blood mononuclear cells extracted from donated patient blood to a combination of vitamin D3 and interleukin 10 to test whether tolerogenic dendritic cells can be generated and have the same functional capacity between donors with and without kidney disease (exposure of PBMC to the uremic environment)

SUMMARY:
The i-KITCaT study aims to harness cellular therapies to favourably alter the immunological response to in AKI in transplantation. Kidney transplantation offers the best survival and quality of life outcomes for patients with end-stage kidney disease but requires life-long immunosuppression. Efforts to increase the donor organ pool means accepting kidneys which have been subjected to medical and surgical factors culminating in acute kidney injury (AKI).

There is no treatment to modify the maladaptive injury process following an AKI insult, and this subjects the new kidney to increased risk of needing dialysis in the first 7 days of transplantation, rejection, and shortened transplant survival.

Tolerogenic dendritic cells (TolDC) are currently used in phase I/II clinical trials and are safe for patients receiving a kidney transplant from the same donor as these cells. These trials focus on transplant tolerance, but we will re-purpose TolDCs to favorably alter the disease course following AKI and limit injury following transplantation.

Furthermore, if the patient's own cells (rather than from a third-party donor) can be used, this avoids supply limitations and potential sensitization risk. We will compare the functional characteristics of TolDC generated from control (healthy) and kidney disease (chronic kidney disease (CKD), dialysis and transplantation).

DETAILED DESCRIPTION:
This observational, cohort study will be conducted at Westmead Hospital

* 3 visits over 24-months per participant.
* each consenting participant will donate 20 - 50ml of peripheral blood per visit.
* recruit n = 20 per study group (control, CKD, dialysis, and transplant).

Aims include:

1. Compare generation of therapeutic grade tolerogenic dendritic cells (TolDC) from peripheral blood mononuclear cells derived from controls (healthy) and patients with kidney disease (CKD, dialysis, or transplantation).
2. Perform testing of TolDC phenotype, tolerogenic capacity and yield.
3. Generate hypothesis for different mechanisms of TolDC function not yet described for further characterisation to support future research

Research plan:

* Peripheral blood mononuclear cells (PBMC) will be isolated from blood by Ficoll gradient and ultrapure magnetic bead sorting.
* PBMC will be tested for purity (other unwanted immune cells) and microbiological contaminants before added to specialized DC media to generate TolDC.
* TolDC will have in depth functional characterization including flow cytometry, cytokine expression, genomic sequencing, and in-vitro testing protocols.
* TolDCs will be co-cultured with human renal cells to test protective capabilities across different AKI stimuli/insults.

This allows selection of ideal PBMC donors to generate functionally desirable TolDC for subsequent use in i-KITCaT studies.

ELIGIBILITY:
Inclusion Criteria:

* able to consent, able to provide blood sample

Exclusion Criteria:

* unable to consent, life-expectancy less than 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study groups
  * Healthy control (eGFR > 90 ml/min/1.73m2 and no known medical issues)
  * Kidney disease with any of the following
  * CKD stage 5 (eGFR < 15 ml/min/1.73m2 from any cause)
  * Dialysis patients (haemodialysis and peritoneal dialysis)
  * Transplant patients (>12-months post-transplant and without prior rejection)
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Tolerogenic dendritic cells | 7 days post ex-vivo culture
  Test flow cytometry, cytokine assays and mixed lymphocyte reaction to show tolerogenic potential of ex-vivo tolerogenic dendritic cells derived from peripheral blood monocytes of donors with and without kidney disease

SECONDARY OUTCOMES:
Transcriptomic differences in tolerogenic dendritic cells derived from healthy and kidney disease donors | 12-months from culture/ex-vivo generation
  transcriptomics (RNA-seq) analysis of differential expression and pathway analysis of tolerogenic dendritic cells derived from both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No